CLINICAL TRIAL: NCT05820789
Title: The Effect of Family Support on Hemodynamic Parameter, Comfort and Anxiety Level in Weaning from Mechanical Ventilation in Cardiovascular Surgery: a Randomized Controlled Study
Brief Title: Family Support Weaning from Mechanical Ventilation in Cardiovascular Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Selda Karaveli Çakır, Assistant professor, Kastamonu University
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-KAEK-146
Record Dates: First submitted 2023-03-14; First posted 2023-04-20 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2024-04

CONDITIONS: Patient Comfort; Anxiety; Patient Satisfaction
Keywords: Weaning; Patient satisfaction; Anxiety; Family support; Cardiac surgery
MeSH Terms: conditions — Anxiety Disorders; Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): When the patient comes intubated from the surgery to the cardiovascular surgery intensive care unit, when they meet the extubation criteria, the patients will be extubated by the healthcare professionals working in the intensive care unit in accordance with the service protocol.Patients in the experimental group will be provided with their relatives and support during weaning from the mechanical ventilator.
  Interventions: Other: Family support
- Control Group (No Intervention): Patient comes intubated from the surgery to the cardiovascular surgery intensive care unit, when they meet the extubation criteria, the patients will be extubated by the healthcare professionals working in the intensive care unit in accordance with the service protocol.

INTERVENTIONS:
Other: Family support — Before the extubation procedure, the patient's relatives will be informed, and the patient will be allowed to enter the intensive care unit, and the patient will be able to express that he is with the patient by holding his hand and talking.
  Other Names: Experimantal group
  Arms: Experimental Group

SUMMARY:
Mechanical ventilation support is used to ensure airway clarity in patients after surgery.If patients are not informed about mechanical ventilation treatment in the pre -operation period, panic, anxiety and comfort may be experienced when they wake up from anesthesia and find them in intensive care under mechanical ventilation with various tubes and equipment. The separation from the mechanical ventilator (MV) covers the patient's mechanical support and the entire process of separation of endotrakeal tube.During the separation of the mechanical ventilator, the support of one of the patient members of the patient may increase the stress and comfort of the patient. Therefore, this research is planned

DETAILED DESCRIPTION:
Intensive care nurses spend a long time with patients and observe them closely. Intensive care nurses in the MV separation process; plays a special and important role. Recently, family support has been used in patient care. An increase in anxiety and comfort levels is observed in patients receiving family support. This study was planned with the aim of supporting the patient by the family member during the separation of the patient from the mechanical ventilator after cardiac surgery and to evaluate the comfort and anxiety level of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research
* To agree to participate in the research verbally and in writing
* To be over the age of 18
* Knowing Turkish
* Not having any psychiatric disease
* No vision, hearing and perception problems
* Receiving mechanical ventilator support after cardiac surgery and being followed in the intensive care unit.

Exclusion Criteria:

* Patients who do not meet the inclusion criteria
* Other patients receiving mechanical ventilator support after surgery in the intensive care unit other than cardiac surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-04-30 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-04-20 (Actual)

PRIMARY OUTCOMES:
State Anxiety | 30 minutes before the weaning procedure.
  State Anxiety Inventory was used to assess state anxiety. The Turkish validity and reliability of the scale were undertaken by Oner and Le Compte . The state anxiety scale composed of 20-items that shows how a person feels at a certain moment and under certain conditions. The scale score ranges from 20 to 80, with a high scores indicating high anxiety.
State Anxiety | after 30 minutes the weaning procedure.
  State Anxiety Inventory was used to assess state anxiety. The Turkish validity and reliability of the scale were undertaken by Oner and Le Compte. The state anxiety scale composed of 20-items that shows how a person feels at a certain moment and under certain conditions. The scale score ranges from 20 to 80, with a high scores indicating high anxiety.
Perianesthesia Comfort | on the 1st day after surgery
  This scale was developed by Kolcaba in 2003, and its Turkish validity and reliability were made by Üstündağ and Eti Aslan in 2010. It is used to evaluate the situation of reaching the expected increase in comfort by determining the comfort requirements. The scale consists of 24 items that question the self-concept and feelings of the individual reflecting the general thought process before and after the surgical intervention. The scale score ranges from 24 to 144, with a high scores indicating high comfort.
Patient's systolic blood pressure (mmHg) | 10 minutes before weaning
  before weaning 1
Diastolic blood pressures (mmHg) | 10 minutes before weaning
  before weaning 2
Heart rate (per minute) | 10 miniutes before weaning procedure
  before weaning 3
Oxygen saturation (SpO2) | 10 miniutes before weaning procedure
  before weaning 4
Patient's systolic blood pressure (mmHg) - after weaning 1 | 10 miniutes after weaning procedure
  Patient's systolic blood pressure (mmHg)
Diastolic blood pressures (mmHg) after weaning 2 | 10 miniutes after weaning procedure
  Diastolic blood pressures (mmHg)
Heart rate (per minute) - after weaning 3 | 10 miniutes after weaning procedure
  Heart rate (per minute)
Oxygen saturation (SpO2) - after weaning 4 | 10 miniutes after weaning procedure
  Oxygen saturation (SpO2)

SECONDARY OUTCOMES:
The Visual Analog Scale | 10 minutes after weaning procedure
  A 10-centimeter vertical VAS was used to assess the satisfaction assessment by patients after weaning procedure. The scale score ranges from 0 to 10, with a high scores indicating high satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Selda Karaveli Cakir, Principal Investigator — Kastamonu Universty
Locations (1):
- Kastamonu University, Kastamonu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No